CLINICAL TRIAL: NCT05374538
Title: A Phase 1a/1b Study of Aurora Kinase A Inhibitor VIC-1911 Monotherapy and in Combination With Sotorasib for the Treatment of KRAS G12C-Mutant Non-Small Cell Lung Cancer
Brief Title: VIC-1911 Monotherapy in Combination With Sotorasib for the Treatment of KRAS G12C-Mutant Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Vitrac Therapeutics, LLC (Industry)
Collaborators: Westat (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIC-1911-01
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: KRAS G12C mutation; AURA kinase; VIC-1911; KRAS G12C; sotorasib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Intervention Model Description: Dose Escalation Phase followed by Expansion Phase. A total of 24 subjects are anticipated in Dose Escalation Phase, Cohort 1a. A total of 12 subjects are anticipated in Dose Escalation Phase, Cohort 1b. A total of 29 subjects are anticipated in Expansion Phase, Cohort 2a. A total of 29 subjects are anticipated in Expansion Phase, Cohort 2b. A total of 46 subjects are anticipated in Expansion Phase, Cohort 2c.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Phase, Cohort 1a: VIC-1911 monotherapy (Experimental): Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy will receive VIC-1911 monotherapy.
  Interventions: Drug: VIC-1911
- Dose Escalation Phase, Cohort 1b: VIC-1911 plus sotorasib combination therapy (Experimental): Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy or are naive to KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.
  Only Dose Level 1 was opened and all 3 subjects received sotorasib 960 mg QD PO, VIC-1911 75 mg BID PO.
  Interventions: Drug: VIC-1911; Drug: sotorasib
- Expansion Phase, Cohort 2a: VIC-1911 monotherapy (Experimental): Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy will receive VIC-1911 monotherapy.
  Interventions: Drug: VIC-1911
- Expansion Phase, Cohort 2b: VIC-1911 plus sotorasib combination therapy (Experimental): Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.
  Interventions: Drug: VIC-1911; Drug: sotorasib
- Expansion Phase, Cohort 2c: VIC-1911 plus sotorasib combination therapy (Experimental): Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC naive to KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.
  Interventions: Drug: VIC-1911; Drug: sotorasib

INTERVENTIONS:
Drug: VIC-1911 — VIC-1911 tablets for oral administration
Drug: sotorasib — Sotorasib tablets for oral administration
  Other Names: LUMAKRAS
  Arms: Dose Escalation Phase, Cohort 1b: VIC-1911 plus sotorasib combination therapy; Expansion Phase, Cohort 2b: VIC-1911 plus sotorasib combination therapy; Expansion Phase, Cohort 2c: VIC-1911 plus sotorasib combination therapy

SUMMARY:
This is a Phase 1a/1b study of aurora kinase A inhibitor VIC-1911 administered as monotherapy and in combination with sotorasib for the treatment of locally advanced or metastatic KRAS G12C-mutant non-small cell lung cancer(NSCLC).

DETAILED DESCRIPTION:
Selected subjects will include males and females age ≥18 years; histologically confirmed locally advanced or metastatic KRAS G12C-mutated NSCLC; received at least 1 prior line of cancer therapy with a PD-1 or PD-L1 inhibitor with or without platinum-based chemotherapy; recovered from all acute toxicities (≤ Grade 1) due to prior therapy; adequate renal and hepatic function; and no known history of significant cardiac, hepatic or ocular disease.

Dose Escalation Phase:

Following screening, a total of up to 36 subjects are anticipated to establish the dose limiting toxicity (DLT) and maximum tolerated doses (MTDs) of VIC-1911 monotherapy and VIC-1911 in combination with sotorasib therapy.

Cohort 1a: Subjects who are refractory to or relapsed on prior KRAS G12C inhibitor therapy will receive VIC-1911 monotherapy. Up to 24 subjects are anticipated in this cohort.

Cohort 1b: Subjects who are refractory to or relapsed on prior KRAS G12C inhibitor therapy or are naïve to KRASG12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy. Up to 12 subjects are anticipated in this cohort.

A 3+3 dose escalation schema will be followed to establish the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of VIC-1911 and VIC-1911 plus sotorasib combination. A total of at least 6 subjects will be treated at the MTD in each group before initiating the Expansion Phase.

Expansion Phase:

Following screening, a total of 104 subjects with KRAS G12C-mutated locally advanced or metastatic NSCLC are anticipated to expand the disease treatment settings of VIC-1911 as monotherapy or in combination with sotorasib. VIC-1911 monotherapy and VIC-1911 plus sotorasib combination therapy will be administered orally at the MTDs established during the Dose Escalation Phase.

Cohort 2a: Subjects who are refractory to or relapsed on prior KRAS G12C inhibitor therapy will receive VIC-1911 monotherapy. (n=29)

Cohort 2b: Subjects who are refractory to or relapsed on prior KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.(n=29)

Cohort 2c: Subjects who are naïve to KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy. (n=46)

VIC-1911 and sotorasib will be taken in the fasted state, 1 hour before or 2 hours after a meal.

Subjects who demonstrate clinical benefit (CR, PR or SD) will be allowed to continue therapy with VIC-1911 and sotorasib until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the subject's condition that prevents further study participation.

Disease response will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST v.1.1).

Blood for hematology, coagulation parameters and serum chemistry determinations and urine will be collected, ECGs will be taken and ophthalmologic exams will be conducted during the study.

Blood will be taken for PK assessment of VIC-1911 and PD assessment of circulating tumor DNA biomarker determinations.

Tumor biopsies will be taken from consenting subjects at Screening and on-study for correlative biomarker determinations. Results will be correlated with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Have locally advanced or metastatic histologically or cytologically confirmed NSCLC, KRAS G12C-mutated
3. The presence of a KRAS G12C mutation should be established prior to entry as assessed in a CLIA qualified laboratory. Testing may be done on tumor tissue (archival or fresh) or on ctDNA from blood.
4. Have received at least 1 prior line of cancer therapy with a PD-1 or PD-L1 inhibitor with or without platinum-based chemotherapy (unless subject is not eligible or refuses chemotherapy or PD-1/PD-L1 therapy and have documented progression on all prior cancer therapies
5. Dose Escalation Phase:

   * Cohort 1a: (VIC-1911 monotherapy): Locally advanced or metastatic NSCLC refractory to or relapsed on at least 1 prior cancer therapy as noted above, and relapsed/refractory on KRAS G12C inhibitor therapy as the most recent cancer therapy prior to study
   * Cohort 1b: (VIC-1911 plus sotorasib): Locally advanced or metastatic NSCLC:

     * Refractory to or relapsed on at least 1 prior cancer therapy as noted above, and relapsed/refractory on KRAS G12C inhibitor therapy as the most recent cancer therapy prior to study, or
     * Refractory to or relapsed on at least 1 prior cancer therapy as noted above, and Naïve to KRAS G12C inhibitor therapy
6. Expansion Phase 1b:

   * Cohort 2a: (VIC-1911 monotherapy): Locally advanced or metastatic NSCLC refractory to or relapsed on at least 1 prior cancer therapy as noted above, and relapsed/refractory on KRAS G12C inhibitor therapy as the most recent cancer therapy prior to study
   * Cohort 2b: (VIC-1911 plus sotorasib): Locally advanced or metastatic NSCLC refractory to or relapsed on at least 1 prior cancer therapy as noted above, and relapsed/refractory on KRAS G12C inhibitor therapy as the most recent cancer therapy prior to study
   * Cohort 2c: (VIC-1911 plus sotorasib): Locally advanced or metastatic NSCLC refractory to or relapsed on at least 1 prior cancer therapy as noted above, and naïve to KRAS G12C inhibitor therapy
7. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
8. Have discontinued previous treatments for cancer, except for sotorasib for subjects to receive VIC-1911 plus sotorasib combination treatment, and have resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior cancer treatment, surgery, or radiotherapy to Grade ≤ 1
9. Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2
10. Life expectancy of ≥ 3 months
11. Subjects with brain metastases:

    11.1 KRAS G12C inhibitor naïve: Subjects with clinically stable (i.e., no increase in corticosteroid requirement) asymptomatic brain metastases are allowed without prior local therapy, as long as all lesions are each ≤ 1 cm. Prior local therapy is required (e.g., stereotactic radiosurgery [SRS], stereotactic body radiation therapy [SBRT], or surgery) for any lesion > 1 cm or any lesion that is symptomatic. Subjects must be clinically stable and asymptomatic following local therapy.

    11.2 KRAS G12C inhibitor pretreated: Subjects with clinically stable (i.e., no increase in corticosteroid requirement) asymptomatic brain metastases following prior local therapy (e.g., SRS, SBRT or surgery) are allowed.
12. Adequate hematologic without ongoing transfusion support:

    * Hemoglobin (Hb) ≥ 8 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9 cells/L
    * Platelets ≥ 75 x 10^9 cells/L
13. Adequate renal and hepatic function:

    * Calculated creatinine clearance ≥ 50 mL/minute x 1.73 m2 per the Cockcroft-Gault formula
    * Total bilirubin ≤ 1.5 times the ULN, unless due to Gilbert's disease, or < 3 times the ULN for subjects with liver metastases
    * ALT/AST ≤ 2 times the ULN, or < 3 times the ULN for subjects with liver metastases
14. Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy throughout the study and for 28 days after the completion of study treatment.
15. Ability to proved written informed consent

Exclusion Criteria:

1. Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV
2. QT interval corrected for rate (QTc) > 480 msec on the ECG obtained at Screening using Fridericia method for QTc calculation
3. Medications that are inhibitors or inducers of UDP-glucuronosyltransferases (UGTs) are prohibited in the Dose Escalation Phase
4. History of corneal epithelial cysts or other ocular events leading to blurred vision, or has medically relevant abnormalities identified on screening ophthalmologic examination
5. Symptomatic pneumonitis/interstitial lung disease requiring medical intervention
6. Symptomatic central nervous system metastasis
7. Leptomeningeal carcinomatosis
8. Inability to swallow oral medication
9. Gastrointestinal conditions that could impair absorption or tolerance of study drugs
10. Current hematologic malignancies
11. Second, active primary solid tumor malignancy that, in the judgement of the Investigator or Sponsor Medical Monitor, may affect the interpretation of results, with the exception of carcinoma in situ of any origin, non-muscle invasive bladder cancer, and Gleason < 3+3 prostate cancer
12. Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment within the last week prior to study treatment
13. Other active infection requiring IV antibiotic usage within the last week prior to study treatment
14. Unable to tolerate marketed dose of KRAS G12C inhibitor on prior therapy for subjects to be enrolled in combination VIC-1911 plus sotorasib treatment cohorts. Alternatively, these subjects may be able to enroll in the VIC-1911 monotherapy treatment cohort, upon discussion with the Medical Monitor and Study Chair.
15. Previous MEK or EGFR inhibitor therapy
16. Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
17. Receipt of an investigational product on a clinical trial within 5 elimination half-lives or within 28 days, whichever is shorter, prior to C1D1 on this study, or currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
18. Previously completed or withdrawn from any other study investigating an aurora kinase A inhibitor
19. Known hypersensitivity to VIC-1911 or its components
20. If female, pregnant, breast-feeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2023-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Goldberg, MD, MPH, Study Chair — Yale Cancer Center, Yale University; Linda J Paradiso, DVM, Study Director — Vitrac Therapeutics, LLC
Locations (5):
- United States (5):
  - University of California Davis, Sacramento, California
  - Yale Cancer Center, North Haven, Connecticut
  - Emory University Winship Cancer Center, Atlanta, Georgia
  - University of Maryland Cancer Center, Baltimore, Maryland
  - New York University Langone Health Perlmutter Cancer Cancer, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy: Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy or are naive to KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.
  VIC-1911: VIC-1911 tablets for oral administration
  sotorasib: Sotorasib tablets for oral administration
  Only Dose Level 1 was opened and all 3 subjects received sotorasib 960 mg QD PO, VIC-1911 75 mg BID PO.
Period: Overall Study
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the same for each group enrolled in the study. Subjects were enrolled only in Cohort 1b.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy | Total
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 0 | 0 | 0 | 2
  >=65 years | 0 | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 60.3 [46 to 74] |  |  |  | 60.3 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 |  |  |  | 2
  Male |  | 1 |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  |  |  | 0
  Not Hispanic or Latino |  | 2 |  |  |  | 2
  Unknown or Not Reported |  | 1 |  |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  |  |  | 0
  Asian |  | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  |  |  | 0
  Black or African American |  | 0 |  |  |  | 0
  White |  | 1 |  |  |  | 1
  More than one race |  | 0 |  |  |  | 0
  Unknown or Not Reported |  | 2 |  |  |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 3 |  |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Safety and tolerability assessed by adverse events(AEs) and serious adverse events (SAEs)
Time Frame: 9 months
Population: No subjects were treated in the Dose Escalation Phase, Cohort 1a. The Expansion Phase did not open.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
Participants | 0 | 3 | 0 | 0 | 0

2. Secondary Outcome: Objective Response Rate
Description: Proportion of subjects with objective responses (complete response [CR] + partial response [PR]) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
Time Frame: Assessed at the end of Cycle 2 and every 2 cycles thereafter up to 8 months. Each cycle is 28 days.
Population: No subjects were treated in the Dose Escalation Phase, Cohort 1a. The Expansion Phase did not open.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of Response
Description: Length of time from first evidence of objective response (complete response [CR] or partial response [PR]) to the first objective evidence of disease progression
Time Frame: Assessed at the end of Cycle 2 and every 2 cycles thereafter up to 8 months. Each cycle is 28 days.
Population: No data displayed because Outcome Measure had zero participants with CR or PR.
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Response
Description: Length of time from the date of first dose of study drug to the first evidence of objective response (CR,PR)
Time Frame: Assessed at the end of Cycle 2 and every 2 cycles thereafter up to 8 months. Each cycle is 28 days.
Population: No data displayed because Outcome Measure had zero participants with CR or PR.
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Disease Control Rate
Description: Proportion of subjects with best response of CR, PR or stable disease (SD)
Time Frame: Assessed at the end of Cycle 2 and every 2 cycles thereafter up to 8 months. Each cycle is 28 days.
Population: No data displayed because Outcome Measure had zero participants with CR, PR or SD.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
Participants |  | 0 |  |  |

6. Secondary Outcome: Progression-Free Survival
Description: Length of time from the date of first dose of study drug to the first evidence of disease progression or death, whichever is earlier
Time Frame: Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier, assessed up to 9 months
Population: No subjects were treated in the Dose Escalation Phase, Cohort 1a. The Expansion Phase did not open.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
days |  | 47 [35 to 61] |  |  |

7. Secondary Outcome: Overall Survival
Description: Length of time from the date of first dose of study drug to date of death from any cause
Time Frame: Assessed from the date of the first dose of study drug to date of death from any cause, assessed up to 9 months
Population: No subjects were treated in the Dose Escalation Phase, Cohort 1a. Death dates reported for 2 of 3 subjects in Cohort 1b. The Expansion Phase did not open.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
days |  | 86 [47 to 125] |  |  |

8. Other Pre Specified Outcome: Mean Plasma Concentrations of VIC-1911 Alone and in Combination With Sotorasib
Description: Mean plasma concentrations of VIC-1911 will be determined and summarized by dose group.
Time Frame: Was to be assessed C1D1; C1D15; C2D1; C4D1; C6D1 (each cycle is 28 days). The study terminated early with only 3 subjects analyzed C1D1 and 2 subjects analyzed C1D15.
Population: No subjects were treated in the Dose Escalation Phase, Cohort 1a. The Expansion Phase did not open.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
ng/mL
  C1D1 |  | 2190 (2090) |  |  |
  C1D15: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  C1D15 |  | 2120 (0) |  |  |

9. Other Pre Specified Outcome: Circulating Tumor DNA (ctDNA) in Plasma (Pharmacodynamic Endpoint)
Description: Changes from baseline will be determined, summarized by dose group and correlated with clinical outcome
Time Frame: Cycle 1 Day 1 pre-dose and at progression of disease
Population: No data displayed because circulating tumor DNA was not collected for this Outcome Measure for any participant.
Groups:
- Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy: Subjects with locally advanced or metastatic KRAS G12C-mutated NSCLC refractory to or relapsed on prior KRASG12C inhibitor therapy or are naive to KRAS G12C inhibitor therapy will receive VIC-1911 plus sotorasib combination therapy.
  VIC-1911: VIC-1911 tablets for oral administration
  sotorasib: Sotorasib tablets for oral administration
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Tumor Biopsies for Biomarker Assessment (Pharmacodynamic Endpoint)
Description: Changes from baseline will be determined, summarized by dose group and correlated with clinical outcome
Time Frame: Pre-study, Cycle 3 Day 1, and at progression of disease
Population: No data displayed because tumor biopsies for this Outcome Measure were not collected for any participant.
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Effect of de Novo Versus Acquired Resistance to KRASG12C Inhibitor Therapy, in Subjects Refractory to or Relapsed on Prior KRAS G12C Inhibitor Therapy
Description: The effect of prior KRAS G12C de novo resistance (KRAS G12C inhibitor treatment ≤ 3 months) versus KRAS G12C acquired resistance (KRAS G12C inhibitor treatment > 3 months) on clinical outcome
Time Frame: 42 months
Population: No data displayed because Outcome Measure had zero participants with clinical outcome CR, PR or SD.
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: No subjects were treated in the Dose Escalation Phase, Cohort 1a. The Expansion Phase did not open.
Arm/Group | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/3 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/3 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy (N=0) | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy (N=3) | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy (N=0) | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy (N=0) | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy (N=0)
Constipation (Gastrointestinal disorders) | NA | 1 (1) | NA | NA | NA
Pneumonia (Infections and infestations) | NA | 1 (1) | NA | NA | NA
Embolism (Vascular disorders) | NA | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase, Cohort 1a: VIC-1911 Monotherapy (N=0) | Dose Escalation Phase, Cohort 1b: VIC-1911 Plus Sotorasib Combination Therapy (N=3) | Expansion Phase, Cohort 2a: VIC-1911 Monotherapy (N=0) | Expansion Phase, Cohort 2b: VIC-1911 Plus Sotorasib Combination Therapy (N=0) | Expansion Phase, Cohort 2c: VIC-1911 Plus Sotorasib Combination Therapy (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema, peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Noncardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalized ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to subsequent approval of additional KRAS G12C inhibitor therapies since this study was initiated, providing clinicians with more choices for treatment of subjects with KRAS G12C-mutant NSCLC. Thus, no formal efficacy analyses, and no pharmacodynamic determinations, were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT05374538/Prot_SAP_000.pdf